CLINICAL TRIAL: NCT00612001
Title: Phase I Study of Glioma-Associated Antigen (GAA) Peptide-pulsed Dendritic Cell Vaccination in Malignant Glioma Patients
Brief Title: Vaccine Therapy in Treating Patients With Malignant Glioma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000585166; R01CA112358 (NIH); UCLA-06-01-052
Record Dates: First submitted 2008-02-08; First posted 2008-02-11 (Estimated); Last update posted 2015-10-05 (Estimated); Status verified 2013-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult anaplastic astrocytoma; adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma; adult anaplastic oligodendroglioma; recurrent adult brain tumor; adult mixed glioma
MeSH Terms: conditions — Central Nervous System Neoplasms; Astrocytoma; Glioblastoma; Gliosarcoma; Oligodendroglioma; Brain Neoplasms; Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- dendritic cell vaccine (Experimental)
  Interventions: Biological: glioma-associated antigen peptide-pulsed autologous dendritic cell vaccine

INTERVENTIONS:
Biological: glioma-associated antigen peptide-pulsed autologous dendritic cell vaccine

SUMMARY:
RATIONALE: Vaccines made from peptides and a person's dendritic cells may help the body build an effective immune response to kill tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in treating patients with malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the dose-limiting toxicity and maximum tolerated dose of autologous dendritic cells pulsed with synthetic glioma-associated antigen (GAA) peptides in patients with malignant gliomas.
* Determine survival, tumor progression, and cellular immune response in patients treated with this regimen.

OUTLINE: Patients undergo leukapheresis for the collection of peripheral blood mononuclear cells (PBMC). Autologous dendritic cells (DC) are prepared from autologous PBMC exposed to sargramostim (GM-CSF) and interleukin-4 (IL-4), matured with a cytokine cocktail, and pulsed with synthetic glioma-associated antigen (GAA) peptides. Cohorts of patients receive escalating doses of GAA peptide-pulsed autologous dendritic cell vaccine until the maximum tolerated dose is determined.

After completion of study treatment, patients are followed every 2 months for 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of 1 of the following malignant gliomas:
* Anaplastic astrocytoma
* Glioblastoma multiforme
* Oligodendroglioma
* Oligoastrocytoma
* WHO grade III or IV disease
* Newly diagnosed or recurrent disease
* Bidimensionally measurable disease by contrast-enhancing MRI
* Surgically accessible tumor for which resection is indicated
* Previously treated with or planning to undergo treatment with conventional external beam radiotherapy
* HLA-A*201 positive
* Karnofsky performance status 60-100%
* Life expectancy ≥ 8 weeks
* Hemoglobin ≥ 10 g/dL
* Absolute granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* SGOT and SGPT ≤ 2 times normal
* Alkaline phosphatase ≤ 2 times normal
* Bilirubin ≤ 1.5 mg/dL
* BUN ≤ 1.5 times normal OR creatinine ≤ 1.5 times normal
* Negative pregnancy test
* Fertile patients must use effective contraception
* Hepatitis B negative
* Hepatitis C negative
* HIV negative
* Syphilis serology negative
* Afebrile

Exclusion Criteria:

* active infection
* immunodeficiency
* autoimmune disease that may be exacerbated by immunotherapy, including any of the following:
* Rheumatoid arthritis
* Systemic lupus erythematosus
* Vasculitis
* Polymyositis-dermatomyositis
* Scleroderma
* Multiple sclerosis
* Juvenile-onset insulin-dependent diabetes
* allergy to study agents
* underlying condition that would contraindicate study therapy
* concurrent severe or unstable medical condition that would preclude giving informed consent
* psychiatric condition that would preclude study participation or giving informed consent
* other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, localized prostate cancer, or carcinoma in situ of the cervix
* prior chemotherapy (6 weeks for nitrosoureas) within last 4 weeks of starting treatment
* concurrent corticosteroids within 2 weeks prior to treatment
* radiotherapy within 2 weeks prior to treatment
* systemic antibiotics within 72 hours prior to treatment
* prior organ allograft
* antihistamine therapy within 5 days before or after administration of study vaccine
* chemotherapy during and for 4 weeks after administration of study vaccine
* adjuvant therapy during and for 4 weeks after administration of study vaccine
* other concurrent investigational agents

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-05; Primary Completion 2011-01 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Dose-limiting toxicity and maximum tolerated dose of autologous dendritic cells pulsed with synthetic glioma-associated antigen (GAA) peptides | 3 months
Survival | 1 year
Tumor progression | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Linda M. Liau, MD, PhD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (1):
- Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California, United States

REFERENCES:
- [Derived] Prins RM, Wang X, Soto H, Young E, Lisiero DN, Fong B, Everson R, Yong WH, Lai A, Li G, Cloughesy TF, Liau LM. Comparison of glioma-associated antigen peptide-loaded versus autologous tumor lysate-loaded dendritic cell vaccination in malignant glioma patients. J Immunother. 2013 Feb;36(2):152-7. doi: 10.1097/CJI.0b013e3182811ae4. PMID 23377664